CLINICAL TRIAL: NCT02075853
Title: Outcomes of the Evans Calcaneal Lengthening Based on Bone Grafting Material
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0531
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; Pes Planus
Keywords: Cerebral palsy; Pes planus; Calcaneal lengthening
MeSH Terms: conditions — Cerebral Palsy; Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Bovine Xenograft: Patients in this group received a bovine xenograft in their Evans calcaneal lengthening procedure. Up until April 2014, patients were randomized into receiving the bovine graft or allograft. However, the bovine xenograft will no longer be manufactured, so no future patients will receive the bovine xenograft during the procedure.
- Iliac Crest Allograft: Patients in this group received an iliac crest cadaver allograft (bicortical or tricortical) in their Evans calcaneal lengthening procedure. Up until April 2014, patients were randomized into receiving the bovine graft or allograft. However, the bovine xenograft will no longer be manufactured, so all future patients will receive the allograft during the procedure.

SUMMARY:
The Evans calcaneal lengthening is a common surgical correction used for children with spastic cerebral palsy (CP) and painful flat feet. This procedure involves the insertion of a trapezoidal bone graft into the calcaneus bone. Both autograft and allografting materials have been used for this procedure, but both types of grafting materials have associated limitations. Autologous grafting materials, which are harvested from the iliac crest at the time of surgery, are associated with high rates of prolonged donor site pain. There is limited bone available from the iliac crest. For this reason autologous bone grafts are not commonly used for the Evan's procedure. Cadaver allografting materials are variable in their mechanical and geometric properties. Recently, xenografting materials have been developed that have consistent mechanical properties and are available in a larger size that is formed to fit the individual patient intraoperatively. The purpose of this study is to evaluate the long term outcomes of the procedure with the different graft options. Another purpose is to compare the difference in surgical correction obtained with the cadaver allograft and the xenografting materials. This study will also observe and evaluate a wide range of outcome variables that encompass multiple levels of patient care, from clinical observation to parent and patient satisfaction, and compare these with the observed changes in the radiographic and plantar pressure parameters of the foot. This data will be evaluated pre to post surgery and for two years of follow-up time. The aim is to uncover the characteristics of collapse observed with the two different grafting materials.

DETAILED DESCRIPTION:
Primary Outcome Measures:

1. Measurement on radiographs of distance between heme clips located in calcaneous bone of the foot. Within the patient's own calcaneous bone, a heme clip will be placed on each side of the osteotomy. From radiographs, the amount of collapse will be determined by measuring the distance from one heme clip to the other. Changes in the distance between the clips indicate collapse of the graft.
2. Radiographic measurements of weight bearing feet of the bovine xenograft group and iliac crest allograft group (tricortical and bicortical), pre-operatively and post-operatively.

   1. Lateral Radiographs: Talocalcaneal angle, Talo first metatarsal angle, Talo horizontal angle, and Calcaneal pitch
   2. Anterior-Posterior Radiographs: Talocalcaneal angle, Talo first metatarsal angle, and Talonavicular coverage
3. Comparison of ligamentous laxity between the two grafting material groups, as measured by the Beighton measurements at patient's pre-operative orthopaedic clinical appointment.

Secondary Outcome Measures:

1. Plantar pressures values of interest are of six segments: medial heel, lateral heel, medial midfoot, lateral midfoot, first metatarsal and second metatarsal. The center of pressure index, total contact area, mean pressure, peak pressure, and pressure time intervals will also be collected and assessed to determine pressure distribution of the foot.

Tertiary Outcome Measures:

1. Health related quality of life assessments between the two groups, pre-operative and post-operative as measured by the Pediatric Orthopaedic Data Collection Instrument (PODCI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic CP or similar neuromuscular disorder
* Surgical correction of pes planovalgus, through the Evans calcaneal lengthening
* Age 4-18 years old
* Gross Motor Function Classification System (GMFCS) 1-4
* Children who are ambulatory or non-ambulatory and able to stand for plantar pressures
* Children who have or will have a first metatarsal osteotomy at the foot

Exclusion Criteria:

* Concomitant bony surgical procedures at the foot either before or concomitantly with the Evans procedure
* Gross Motor Function Classification System (GMFCS) level of 5

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children receiving an Evans calcaneal lengthening procedure at Children's Hospital Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Change in the amount of collapse | Pre-operatively (3-12 months), 6 weeks, 6 months, and 1 and 2 years post-operatively
  Measurement on radiographs of distance between heme clips located in calcaneous bone of the foot. Within the patient's own calcaneous bone, a heme clip will be placed on each side of the osteotomy. From post-operative radiographs, the amount of collapse will be determined by measuring the distance from one heme clip to the other. Post-operative changes in the distance between the clips from the first radiograph after surgery (used as a baseline, usually 6 weeks after surgery) indicate collapse of the graft.

SECONDARY OUTCOMES:
Change in Plantar pressures | Pre-operatively (3-12 months), then 1 and 2 years post-operatively
  Plantar pressures values of interest are of six segments: medial heel, lateral heel, medial midfoot, lateral midfoot, first metatarsal and second metatarsal. The center of pressure index, total contact area, mean pressure, peak pressure, and pressure time intervals will also be collected and assessed to determine pressure distribution of the foot. Change from baseline (pre-operative measurements) will be evaluated up to 2 years post-operatively. The pre-operative plantar pressures must be within a year of the surgery.

OTHER OUTCOMES:
Change in Health related quality of life | Pre-operativey (3-12 months), then at 6 months, 1 and 2 years post-operatively
  Health related quality of life assessments between the two groups, preoperative and post-operative as measured by the Pediatric Orthopaedic Data Collection Instrument (PODCI) questionnaire. Pre-operative assessments must be within a year before surgery, and post-operative assessments will be conducted up to 2 years post-operatively to compare the changes from baseline (from pre-operative assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Chang, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States